CLINICAL TRIAL: NCT02988791
Title: Randomized Clinical Trial to Evaluate the Efficacy of Bifidobacterium in the Treatment of Infantile Colic (IC)
Brief Title: Evaluation of a Probiotic (Bifidobacterium in the Treatment of Infantile Colic (IC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: SOFAR S.p.A. (Industry)
Responsible Party: Principal Investigator, Roberto Berni Canani, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250
Record Dates: First submitted 2016-11-14; First posted 2016-12-09 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Probiotic (Bifidobacterium) (Experimental): Active, Bifidobacterium BB12
  Interventions: Dietary Supplement: probiotic (BIfidobacterium, BB-12®)
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: probiotic (BIfidobacterium, BB-12®) — probiotic (Bifidobacterium, BB-12®)
  Arms: Probiotic (Bifidobacterium)
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Infantile colic (IC) criteria includes all of the following in subjects aged ≤ 4 months: paroxysms of irritability, fussing, or crying that start and stop without obvious cause; episodes lasting 3 or more hours per day and occurring at least 3 days per week for at least 1 week; and no failure to thrive. The condition is very common in the first 4 months of life (10-30 % of infants) with a peak prevalence at 6-8 weeks and is characterized by excessive and inconsolable crying without an identifiable cause. Infantile colic cause considerable stress for the baby and the family, huge medical expenses (the IC cause 10-20 % of all pediatric visits in the first 4 months of life) and frequent formula changes.

The pathophysiology of IC is still poorly defined, but differences in gut microbiota composition seem to be involved. In particular, differences in the number and species of Lactobacilli spp, Klebsiella spp and Escherichia coli spp have been demonstrated in subjects with IC, and it has been postulated that these alterations could be responsible for an abnormal gas production within gut lumen resulting in distension and abdominal pain. These findings suggest the potential role of probiotics as preventive and therapeutic strategy for the IC.

ELIGIBILITY:
Inclusion Criteria:

* exclusively breastfed healthy infants of both sex, aged ≤ 7 weeks;
* Diagnosis of IC according to Rome III criteria
* Written informed consent of the parent/tutor

Exclusion Criteria:

* Birth weight<2500 g
* Gestational age<37 weeks
* APGAR 5 minutes <7
* Formula feeding
* Abnormal body growth/loss of weight (<100 g/weeks from birth to the last reported weight)
* Neurological diseases
* Known or suspected food allergy
* Gastroesophageal reflux disease
* Use of substances that alter gut microbiota (pre/pro/synbiotic, antibiotics, gastric acidity inhibitors) or any anti-colic drug in the last 2 weeks prior the enrollment
* History of fever and/or infectious diseases in the last 2 weeks prior the enrollment
* Ongoing systemic infections
* History of congenital infections
* Chronic intestinal diseases (cystic fibrosis or other forms of pancreatic insufficiency primitive)
* Malformation of the gastrointestinal (such as esophageal atresia, intestinal atresia, short bowel syndrome, malrotation), urinary or respiratory tract
* Metabolic diseases
* Genetic diseases and chromosomal abnormalities
* Primary or secondary immunodeficiencies
* Not sufficient reliability or presence of conditions that may result in non-compliance/adherence of the patient to the Protocol
* Previous participation in this study

Ages: 1 Week to 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
mean daily crying duration | up to 28 days
  reduction of ≥50% of mean daily crying duration

SECONDARY OUTCOMES:
number of regurgitation | up to 28 days
Evaluation of the gut microbiota modifications | up to 28 days
  Stool sample
fecal production of peptides from innate immune system | up to 28 days
  Stool sample
fecal short chain fatty acids production | 28 days
  Stool sample
evacuative frequency | up to 28 days
consistency of the fecal mass | up to 28 days
  assessed by means of Bristol score
number of crying episode | up to 28 days
sleep | up to 28 days
  duration of sleep

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy